CLINICAL TRIAL: NCT01822093
Title: Phase I/II Study Investigating the Safety of ADV Specific T Cells in High-risk Paediatric Patients Post Allo-HSCT to Treat ADV Reactivation
Brief Title: Safety Study of ADV-specific T-cells in Paediatric Patients Post Allo-HSCT
Acronym: ASPIRE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cell Medica Ltd (Industry)
Collaborators: Technology Strategy Board, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM-2011-02
Record Dates: First submitted 2013-02-11; First posted 2013-04-02 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: ADV Infection Post Allo-HSCT

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cytovir-ADV (Experimental): Adenovirus-specific T-cells
  Interventions: Biological: Cytovir-ADV

INTERVENTIONS:
Biological: Cytovir-ADV — A single dose 1x10e4 CD3+ T cells/kg patient weight of Cytovir ADV is prescribed to patients on exhibiting two consecutive PCR positive Adenovirus viraemia results > 1000 copies/ml. Patients are followed up by continued monitoring of Adenovirus viraemia results. If patients exhibit uncontrolled ADV viraemia at ≥ 4 weeks following the first cell dose, they will be prescribed a second cell dose of 10e5 CD3+ T cell/kg. Patients will be monitored for 6 months following infusion of Cytovir ADV.
  This is a feasibility/pilot study and has no control group
  Other Names: Adenovirus-specific T-cells

SUMMARY:
Human Adenovirus-specific T-cells can persist and augment impaired adenovirus immune response post allogeneic haematopoietic stem cell transplant, and reduce the requirement for antiviral therapy without toxicity or increasing the occurrence of Graft Versus Host Disease. This is a Phase I/IIa open-label safety study, assessing the effects of administering adenovirus-specific T-cells (Cytovir ADV) to paediatric patients post haematopoietic stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

Patients:

1. Age 16 years or younger
2. Scheduled to undergo an allogeneic HSCT with an unrelated donor, mismatched unrelated donor, mismatched family donor or haplo identical donor
3. The subject (or legally acceptable representative) must give informed consent (and assent for subjects ≥ 12 years). All subjects will have a parent or guardian provide informed consent and the subject will provide witnessed verbal assent
4. Negative serology for HIV 1 + 2, HepB, HepC, Syphilis, hCG.

Donors

1. Meets requirements of Directive 2004/23/EC as amended and the UK statutory instruments pursuant therein
2. Negative serology for HIV 1 + 2, HepB, HepC, Syphilis, hCG
3. Passed medical assessment for stem cell donation
4. HdADV seropositive
5. Signed informed consent
6. Age 16 years or older

Exclusion Criteria:

Patients

1. Pregnant or lactating females
2. Co-existing medical problems that would place the patient at significant risk of death due to GVHD or its sequelae
3. Human Immunodeficiency Virus (HIV) infection

Donors

1. Pregnant or lactating females
2. (assessed prior to apheresis) Platelets < 50x109/L

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2012-12; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Number of subjects with new onset GVHD | 180 days
number of subjects developing NCI Grade 3-4 adverse events | 180 days

SECONDARY OUTCOMES:
Number of reported Serious Adverse Events (SAEs), Suspected Unexpected Serious Adverse Reactions (SUSARs) and Suspected Expected Serious Adverse Reactions (SESARs) | 180 days
Number of detectable HAdV-specific T-cells in vivo at each time point | 180 days
Requirement for second infusion of HAdV-specific T-cells | 180 days
Number of treatment days with antiviral drugs | 180 days
Number of treatment days with other anti-infective drugs | 180 days
Number of in-hospital days during 6 month post-infusion period | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Waseem Qasim, Principal Investigator — Institute of Child Health, London
Locations (3):
- United Kingdom (3):
  - Great Ormond Street Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Royal Victoria Infirmary, Newcastle